CLINICAL TRIAL: NCT06075017
Title: Comparison of Biofilm Accumulation on the Surface of Zirconia Versus Titanium Implants. Randomized Controlled Pilot Clinical Trial
Brief Title: Biofilm Accumulation in Zirconia vs. Titanium Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 109-190723
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-12

CONDITIONS: Implant Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zirconia (Experimental): Two-piece zirconia dental implant will be placed to replace a single missing tooth.
  Interventions: Procedure: dental implant placement
- Titanium (Active Comparator): Two-piece titanium dental implant will be placed to replace a single missing tooth.
  Interventions: Procedure: dental implant placement

INTERVENTIONS:
Procedure: dental implant placement — Comparing the amount and type of biofilm on zirconia vs. titanium implants
  Other Names: Titanium dental implants

SUMMARY:
The aim of this randomized clinical trial is to compare the amount and type of biofilm formed on the surface of zirconia implants compared to titanium implants.

A pilot randomized clinical trial will be conducted in which 15 zirconia and 15 titanium single implants will be placed in different patients and the amount of total biofilm and different bacterial species will be evaluated at 3, 6 and 12 months after placement, in addition to bleeding on probing, plaque index, amount of keratinized gingiva, marginal bone loss and patient satisfaction. The Shapiro-Wilk normality test will be performed to determine whether each group follows a normal distribution. Once the distribution of the samples has been verified, we will proceed to apply a parametric test of repeated measures ANOVA or mixed ANOVA with Bonferroni correction, in order to observe what changes exist in the variables to be studied and if these will be statistically significant, establishing a significance level of P<0.05. If the distribution does not comply with normality, the nonparametric Friedman test will be performed.

DETAILED DESCRIPTION:
Study design:

The present protocol is designed as a randomized controlled clinical trial. The set of procedures of the present clinical trial will be carried out in the Master of Oral Surgery and Implantology of the Faculty of Dentistry of the Complutense University of Madrid (Spain). This study will be carried out in accordance with the principles established by the Declaration of Helsinki and will be conducted under the approval of the Clinical Trials Committee of the Hospital Clínico San Carlos of Madrid.

The selection of subjects with indication for osseointegrated implant placement will be based on a previous oral and radiological examination by means of a periapical radiograph and a panoramic radiograph and/or Cone Beam Computed Tomography , together with the completion of a clinical questionnaire.

For implant placement, a linear incision of the edentulous ridge and an intrasulcular incision of the adjacent teeth will be made using a #15 scalpel blade and a #3 Bard Parker scalpel handle. Once this is done, a full-thickness flap will be raised and the alveolar ridge will be reamed, following the manufacturer's indications, to place a titanium implant (Phibo® Aurea Evolution) of adequate dimensions in the control group or a zirconia implant (Z system®) in the test group, checking that there is an adequate insertion torque of 30Ncm or more and a cover screw will be placed. Once the implant is in place, simple stitches with supramid monofilament 4/0 suture (Proclinic®) will be placed until the wound is closed. Finally, antibiotic treatment (Amoxicillin 750mg/8hours/7 days), analgesic and anti-inflammatory (Dexketoprofen 25mg/8hours/5 days and Metamizole 575mg/8hours/if pain persists) will be prescribed to all patients. Physical anti-inflammatory measures (intermittent local icing for at least 30 minutes) and salt and water rinses 3 times a day for 7 days will be prescribed. Three months after implant placement in the mandible and four months in the maxilla, the final screw-retained metal-ceramic crown will be loaded with a transepithelial abutment made of titanium for titanium implants or zirconia for zirconia implants.

Study visits In both groups, paper-tip samples will be taken from the peri-implant sulcus before the placement of the final crown ("basal" visit), at 6 months (visit 2) and 1 year (visit 3), to perform a culture of the type and quantity of bacteria present in the placed implants. The survival of the placed implants, the probing depth of the implants, the bleeding on probing of the implants, the plaque index of the implants and the amount of keratinized gingiva from the midpoint of the vestibular gingival margin to the mucogingival line on the day of crown placement will also be evaluated at 6 and 12 months. Finally, after final crown placement, a periapical radiograph with parallelizer will be taken and repeated at 6 and 12 months to evaluate marginal bone loss, mesial and distal to the implant, using Vistasoft® 3.0.22/2023 software, calibrating the image with the length of the implant, since its dimension will be known.

Sample size:

Because the data to be analyzed do not coincide with data reflected in studies analyzing biofilm accumulation on the surface of zirconia versus titanium implants, we will conduct a pilot study with 30 subjects (15 in each group), so as to ensure robustness of the results. Based on these results, means and variances, we will perform a sample size calculation for future more comprehensive investigations.

Randomization:

The randomization of this clinical trial will be carried out before the start of the study using the block method, to ensure a periodic balance in the number of subjects assigned to each intervention group and to guarantee the equality of the sample size in the two groups being compared, for this purpose 6 blocks of 5 subjects each will be used.

The computer application IBM® SPSS Statistics version 28.0.1.1 and the macro RNDSEQ will be used for this purpose.

The sequence of intervention assignment will be ignored by the data examiner and by the surgeon, only the data monitor (F.P.G), who will deliver a sealed envelope to the surgeon on the day of implant placement and will have no contact with the patients, will know it.

calibration:In order for the measurements of the secondary variable probing depth, amount of keratinized gingiva and marginal bone loss to be valid and reproducible, an examiner (S.B.B) will take 5 samples on the same patient from a single implant comparing the results by intraclass correlation coefficient using the computer application IBM® SPSS Statistics version 28.0.1.1.

Statistical analysis:

Mean values and standard deviations will be determined for each of the parameters in the test and control group. For the statistical analysis of the results obtained, the computer application IBM® SPSS Statistics version 28.0.1.1 will be used. The Shapiro-Wilk normality test will be performed to determine whether each group follows a normalized distribution, since the sample is smaller than 50 subjects. Once the normalized distribution of the samples has been verified, a parametric test of repeated measures ANOVA or mixed ANOVA with Bonferroni correction will be applied to observe what changes exist in the variables to be studied and if these will be statistically significant, establishing a significance level of P<0.05. If the distribution does not comply with normality, the nonparametric Friedman test will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes of legal age.
* Patients ASA I, II and III.
* Subsequent to the placement of a single implant.
* Patients who accept the surgery and sign the informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients who cannot attend follow-up appointments after surgery.
* Patients with implants adjacent to the area to be treated.
* Patients with uncontrolled periodontal pathology.
* Systemic pathology that contraindicates the surgical procedure: hepatitis or other infectious diseases, oncological treatment, untreated or uncontrolled systemic pathology: diabetes mellitus, arterial hypertension, osteoporosis, heart failure, valvular heart disease, history of endocarditis, acute myocardial infarction less than 6 months ago, stroke less than 6 months ago, history of venous thromboembolism, arrhythmias, vitamin D deficiency, Parkinson's and Alzheimer's disease, dementia, psychiatric disorders, liver disease, COPD, chronic renal failure, immunosuppressed, autoimmune diseases, inflammatory bowel disease, digestive pathology, phosphocalcium metabolism diseases, hyper- or hypothyroidism, endocrinopathies, celiac disease, collagenosis, etc.
* Pharmacological treatment with anticoagulants, antiaggregants, bisphosphonates, monoclonal antibodies, serotonin reuptake inhibitors, immunosuppressants, corticosteroids, antipsychotics.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
total amount of biofilm | 12 months
  The total amount of biofilm (CFU/ml) and the amount of A. actinomyces (CFU/ml), P. gingivalis (CFU/ml), P. intermedia (CFU/ml), T. forsythia (CFU/ml), P. micra (CFU/ml), F. nucleatum (CFU/ml), C. rectus (CFU/ml), E. corrodens (CFU/ml), Capnocytophaga sp. (CFU/ml), A. odontolyticus (CFU/ml), S. mutans (CFU/ml) and Candidae sp. (CFU/ml) on implants placed prior to crown placement, at 6 months and 1 year after final crown placement, by culturing with two sterile paper tips at the two points of greatest probing for 20 seconds each.

CONTACTS AND LOCATIONS:
Locations (1):
- Complutense University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
quantity and type of biofilm on implants and clinical and biological parameters of implants